CLINICAL TRIAL: NCT03606226
Title: FAMILY Holistic Health: Physical Activity and Dietary Attitudes and Behavioural Patterns of Chinese-speaking Individuals in the Hong Kong Community.
Brief Title: Physical Activity and Dietary Attitudes and Behavioural Patterns in the Hong Kong Community
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2019
Record Dates: First submitted 2018-07-16; First posted 2018-07-30 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Physical Activity; Dietary Habits
MeSH Terms: conditions — Motor Activity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The health benefits of regular physical activity and a healthy diet are well established in literature. Regular physical activity and a healthy diet may reduce the risk of certain non-communicable diseases such as diabetes, heart disease, stroke, and cancer, and contribute to mental health and emotional benefits, as well as social wellbeing.

Despite the health benefits of regular physical activity and healthy diet, most of the Hong Kong people live a sedentary and unhealthy lifestyle and do not meet the WHO's recommendation on physical activity for health and on fruit and vegetables intake.

This study is to examine the physical activity and dietary attitudes and behavioural patterns of the Hong Kong community and provide a clear direction for future health education and awareness projects and campaigns aimed towards improving the general health of the Hong Kong community.

DETAILED DESCRIPTION:
The health benefits of regular physical activity and a healthy diet are well established in health literature. Regular physical activity is positively associated with psychological well-being (Bize, Johnson, & Plotnikoff, 2007), and inversely correlated with various illnesses (Pedersen & Saltin, 2006). Similarly, a healthy diet may reduce the risk of certain non-communicable diseases such as diabetes, heart disease, stroke, and cancer (World Health Organization, 2015a; Centers for Disease Control and Prevention (CDC), 2015), , and can also contribute to mental health and emotional benefits, as well as social well-being (Schooling, 2006).

The consequences of physical inactivity and an unhealthy diet are also well established in the literature, with the World Health Organization (WHO) reporting that physical inactivity and unhealthy diets are two of the four main modifiable behavioural risk factors that contribute to non-communicable diseases such as heart diseases, diabetes, and obesity.

Given the health benefits of regular physical activity and the detrimental effects of physical inactivity, the WHO recommends that children and young people aged 5 - 17 years should perform at least 60 minutes of moderate- or vigorous-intensity physical activity per day, and adults aged 18 years or above should perform at least 150 minutes of moderate-intensity or 75 minutes of vigorous-intensity aerobic physical activity per week. In terms of diet, the WHO recommends that for adults that a daily healthy diet should contain at least 5 servings of fruits and vegetables, no more than 50 g of free sugars, and no more than 5 g of salt.

Despite the health benefits of regular physical activity, most Hong Kong people live a sedentary lifestyle. Many do not meet the World Health Organization targets for physical activity. The Department of Health (2015) reports that only 15.3% of local children aged 5 - 14 years meet the WHO recommendations on physical activity for health, and the 2014 Behavioural Risk Factor Survey indicates that only 37.4% of local adults aged 18 - 64 years meet the WHO recommendations on physical activity for health. Similarly, most Hong Kong people do not adopt a healthy diet, with about four-fifths (79.0%) of adults aged 18 - 64 years failing to meet the WHO's recommendation on fruits and vegetable intake. Only 18.7% of local adults aged 18 - 64 years consume 5 or more servings of fruits and vegetables a day (WHO, 2015b; WHO, 2016).

As the aforementioned figures indicate, members of the Hong Kong community do not meet the WHO recommended physical activity and healthy diet standards. Since these standards of regular physical activity and a healthy diet benefit health and wellbeing and can protect against non-communicable diseases, it is important, in order to improve general health, to improve physical activity and healthy diet practices and patterns in the Hong Kong community.

This study is to examine the Hong Kong people's attitudes and behavioural patterns in relation to physical activity and a healthy diet. Attitude-behaviour gaps may be identified, providing a clear starting point and direction for future health education and awareness projects and campaigns aimed towards improving the general health of the Hong Kong community.

ELIGIBILITY:
Inclusion Criteria:

Community events

* Chinese-speaking;
* Aged 13 - 17 years with a legal guardian present, or aged 18 years and above; and
* Able to complete the questionnaire.

Community workshops

* Chinese-speaking;
* Aged 18 years and above; and
* Able to complete the questionnaire.

Exclusion Criteria:

* Individuals failing to meet the inclusion criteria.

Ages: 13 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Chinese-speaking individuals in the Hong Kong community
Sampling Method: Non-Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Attitude on performing physical activity | baseline
  Attitude on performing physical activity will be assessed by outcome-based physical activity questionaire
Attitude on taking dietary habit | baseline
  Attitude on taking healthy diet will be assessed by outcome-based dietary questionnaire

SECONDARY OUTCOMES:
Behaviour on performing physical activity | baseline
  Behaviour on performing physical activity will be assessed by outcome-based questionnaire
Behaviour on taking healthy diet | baseline
  Behaviour on performing healthy diet will be assessed by outcome-based questionnaire
Behaviour on performing physical activity with family members | baseline
  Behaviour on performing physical activity with family members will be assessed by outcome-based questionnaire
Personal well-being | baseline
  Personal health and happines will be assessed by outcome-based questionnaire
Family well-being | baseline
  Family health, happiness and harmony will be assessed by outcome-based questionnaire
Body composition | baseline
  Body mass Index will be measured by an electronic scale
Physical fitness performance (Handgrip strength) | baseline
  Handgrip strength will be measured by dynamometry
Physical fitness performance (Flexibility) | baseline
  Flexibility will be assessed by Chair sit-and-reach test
Physical fitness performance (Balance) | baseline
  Balance will be assessed by single leg stance test
Physical fitness performance (Muscle strength) | baseline
  Lower limb muscle strength will be assessed by sit and stand test

CONTACTS AND LOCATIONS:
Locations (1):
- The Univeristy of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bize R, Johnson JA, Plotnikoff RC. Physical activity level and health-related quality of life in the general adult population: a systematic review. Prev Med. 2007 Dec;45(6):401-15. doi: 10.1016/j.ypmed.2007.07.017. Epub 2007 Jul 21. PMID 17707498
- [Background] Pedersen BK, Saltin B. Evidence for prescribing exercise as therapy in chronic disease. Scand J Med Sci Sports. 2006 Feb;16 Suppl 1:3-63. doi: 10.1111/j.1600-0838.2006.00520.x. PMID 16451303
- [Background] Schooling CM, Lam TH, Li ZB, Ho SY, Chan WM, Ho KS, Tham MK, Cowling BJ, Leung GM. Obesity, physical activity, and mortality in a prospective chinese elderly cohort. Arch Intern Med. 2006 Jul 24;166(14):1498-504. doi: 10.1001/archinte.166.14.1498. PMID 16864760
- See also: Department of Health. (2015a) Healthy Diet — http://www.change4health.gov.hk/en/healthy_diet/figures/index_t.html
- See also: Department of Health. (2015b) Physical Activity — http://www.change4health.gov.hk/en/physical_activity/figures/index_t.html
- See also: World Health Organization. (2010) Global Recommendations on Physical Activity for Health. — http://apps.who.int/iris/bitstream/10665/44399/1/9789241599979_eng.pdf
- See also: World Health Organization. (2015a) Healthy diet. — http://www.who.int/mediacentre/factsheets/fs394/en/
- See also: World Health Organization. (2015b) Noncommunicable diseases. — http://www.who.int/mediacentre/factsheets/fs355/en/
- See also: World Health Organization. (2016) Benefits of a balanced diet. — http://www.euro.who.int/en/health-topics/disease-prevention/nutrition/a-healthy-lifestyle/benefits-of-a-balanced-diet